CLINICAL TRIAL: NCT05616247
Title: Immediate and Long-term Efficacy of the Expectancy Challenge Alcohol Literacy Curriculum on Reducing Adverse Alcohol Outcomes
Brief Title: Efficacy of the Expectancy Challenge Alcohol Literacy Curriculum on Reducing College Student Alcohol Use and Harms
Acronym: ECALC
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R15AA028909-01A1 (NIH)
Record Dates: First submitted 2022-11-07; First posted 2022-11-15 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2024-05

CONDITIONS: Alcohol Use, Underage; Harmful; Use, Alcohol
Keywords: College Alcohol Use; Expectancies; Expectancy Challenge; Expectancy Challenge Alcohol Literacy Curriculum; Alcohol-Related Harms; Underage Alcohol Use
MeSH Terms: conditions — Underage Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- ECALC (Experimental): Cognitive Behavioral Program to Change Expectancy Processes
  Interventions: Behavioral: ECALC
- ECALC Plus Weekly Boosters (Experimental): Cognitive Behavioral Program to Change Expectancy Processes with Weekly Booster Content Delivered by Mobile Device
  Interventions: Behavioral: ECALC Plus Weekly Boosters
- Control (No Intervention): Control Group Presentation on Body Image

INTERVENTIONS:
Behavioral: ECALC — Expectancy Challenge Alcohol Literacy Curriculum Cognitive Behavioral Intervention
  Arms: ECALC
Behavioral: ECALC Plus Weekly Boosters — Expectancy Challenge Alcohol Literacy Curriculum Cognitive Behavioral Intervention Plus Weekly Booster Content Delivered by Mobile Device
  Arms: ECALC Plus Weekly Boosters

SUMMARY:
The current project uses a web-based program called the Expectancy Challenge Alcohol Literacy Curriculum (ECALC) to reduce alcohol use and associated harms among college students. Participants complete the interactive program in 50 minutes, and then provide daily, real-time data on expectancies and alcohol use for 3 weeks after intervention, and again for one week at 13 and 25 weeks after intervention. One group will also receive biweekly boosters delivered via smart phone to assess their impact on intervention decay over time. It is hypothesized that ECALC effects may decay over time, and that biweekly boosters will prevent this decay. Access to the ECALC is available on request from the principal investigator.

DETAILED DESCRIPTION:
The Expectancy Challenge Alcohol Literacy Curriculum (ECALC) is a 50-minute interactive program, and the only non-experiential expectancy challenge that has been successful in significantly reducing alcohol use and harms among college students. In studies focused on mandated students, fraternity and sorority members, and first year college students, ECALC has produced larger effect sizes than experiential expectancy challenge and all widely used programs. ECALC outcome studies have thus far been limited to four weeks, but the design of ECALC suggests that effects might be sustained for much longer. The primary aim of the proposed project is to conduct an RCT designed to evaluate duration of ECALC effects over the course of 6 months, and to assess the impact of smart phone-delivered boosters on maintenance and enhancement of effects. Participants will be problematic drinking college students recruited from first time in college new students. Students will be randomly assigned to ECALC only, ECALC plus boosters, or assessment only control. Ecological momentary assessment (EMA) will be used to track alcohol use and expectancies for one week at baseline, three weeks post-intervention, and one-week intervals at 3 and 6 months. It is hypothesized that students who complete ECALC will demonstrate immediate changes in alcohol expectancies, and subsequently, this will drive lower alcohol use and lower rates of alcohol-related problems (relative to the assessment only control students). It is also hypothesized that changes in expectancies and reduction in alcohol use may decay over time among students who do not receive boosters, while biweekly boosters will promote maintenance or enhancement of effects. This study allows for the examination of (1) duration of ECALC effects up to 6 months, and (2) the impact of biweekly boosters delivered via smart phones. In addition, use of EMA to collect real time data on expectancies and alcohol use over the course of 6 months will allow us to (3) map potential changes in expectancies in relation to alcohol use during this critical period of transition. If successful, this project will validate the use of ECALC as an efficient and effective program for reducing alcohol use and drinking-related harms.

ELIGIBILITY:
Inclusion Criteria:

* Full-time Fist Year College Student
* AUDIT-C score = 5 or higher (women), 7 or higher (men).
* Fluent English speaker
* Able to consent to participate in research

Exclusion Criteria:

* Not a Student enrolled at University of Central Florida
* Pregnant
* AUDIT score =15 or higher

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2022-09-22 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Alcohol Expectancies Measured Weekly with CEOA | Weeks 1, 2, 3, 4, 13, and 26
  Expected effects of alcohol use measured with self-report survey. The survey is the 38 item Comprehensive Effects of Alcohol Scale (CEOA), a validated measure of alcohol expectancies. Participants complete the CEOA online on their mobile device and enter responses to each item. Scores range from 0 to 114 with higher scores indicating greater expectation of effects of consuming alcohol.
Change from Baseline in Alcohol Use Measured Weekly with Retrospective Self-report Measure | Weeks 1, 2, 3, 4, 13, and 26
  Self-reported alcohol use, quantity and frequency of consumption in standard drink format. Participants complete an online survey on their mobile device and enter the number of standard drinks consumed each day and number of hours spent drinking each day over the previous week.
Change from Baseline in Alcohol-related Harms Measured Weekly with Retrospective Self-report Survey | Weeks 1, 2, 3, 4, 13, and 26
  Self-reported Negative consequences associated with alcohol use measured with self-report survey. Participants complete an online survey on their mobile device. The survey is the Young Adult Alcohol Consequences Questionnaire. A 48-item validated measure with scores ranging from 0 to 67, higher scores indicate more harms.
Change from Baseline in Sociocultural Attitudes Towards Appearance Measured Weekly with Self-report Survey | Weeks 1, 2, 3, 4, 13, and 26
  Attitudes toward personal appearance measured with self-report survey. Participants complete an online survey on their mobile device. The survey is the Sociocultural Attitudes Towards Appearance Questionnaire-4. A 22-item validated measure with scores ranging from 0 to 110, higher scores indicate more sociocultural emphasis on personal appearance and body image.
Change from Baseline in Alcohol Expectancies Measured Daily with Ecological Momentary Assessment (EMA) | Daily for Weeks 1, 2, 3, 4, 13, and 26
  Expected effects of alcohol use measured with 8 item self-report survey. Participants complete an online survey on their mobile device and enter responses to items each day. Scores range from 0 to 24 with higher scores indicating greater expectation of effects of consuming alcohol. Items were selected from the Comprehensive Expected Effects of Alcohol Scale (CEOA).
Change from Baseline in Alcohol Use Measured Daily with Ecological Momentary Assessment (EMA) | Daily for Weeks 1, 2, 3, 4, 13, and 26
  Self-reported alcohol use, quantity and frequency of consumption in standard drink format. Participants complete an online survey on their mobile device and enter the number of standard drinks consumed each day.

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Dunn, Ph.D., Principal Investigator — University of Central Florida
Locations (1):
- University of Central Florida, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Didentified data will be placed in NIH approved data repository (currently https://cos.io/our-products/osf/).
Supporting Information: Study Protocol, SAP
Time Frame: Data available May 01, 2026 Availability indefinite
Access Criteria: Access will be open.